CLINICAL TRIAL: NCT00716768
Title: Randomized Controlled Trial of Laparoscopic Compared to Open Inguinal Hernia Repair in Children Younger Than 3 Years of Age
Brief Title: Trial of Laparoscopic Compared to Open Inguinal Hernia Repair in Children Younger Than 3 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Fizan Abdullah, MD, Associate Professor of Surgery, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00010962
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Inguinal Hernia
Keywords: Laparoscopic; Inguinal Hernia; Infants
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Inguinal Hernia Repair (Active Comparator)
  Interventions: Procedure: Laparoscopic Inguinal Hernia Repair
- Open Inguinal Hernia Repair (Active Comparator)
  Interventions: Procedure: Open Inguinal Hernia Repair

INTERVENTIONS:
Procedure: Laparoscopic Inguinal Hernia Repair — Laparoscopic Inguinal Hernia Repair
  Arms: Laparoscopic Inguinal Hernia Repair
Procedure: Open Inguinal Hernia Repair — Open Inguinal Hernia Repair
  Arms: Open Inguinal Hernia Repair

SUMMARY:
Laparoscopic techniques have been applied widely to the management of various common pediatric surgical diseases. Current evidence lacks sufficient quality to justify the widespread adoption of the laparoscopic approach to the repair of inguinal hernias within children. It is important to critically evaluate the efficiency and the potential risks of these new techniques before they can supplant open techniques as the treatment modality of choice. Numerous large case series of laparoscopic inguinal hernia repair have been reported with average length of stay, complication rates, recurrence rates and pain management scores that mirror those of open inguinal hernia repair. Only one randomized controlled trial has been performed to compare the open versus laparoscopic technique which has not provided answers regarding the potential benefits on young infants. Benefits of an open approach in children includes a shorter operative time, while the laparoscopic procedure is associated with less pain and a better cosmetic result.

This study will compare open versus laparoscopic repairs of inguinal hernias. The primary outcome variable will be total dose of acetaminophen administered postoperatively for pain management. Secondary outcome variables include 1) Incidence of intraoperative complications such as compromise of testicular vessels, perforation of abdominal viscera; 2) Short-term outcomes such as operative time, rate of conversion from open to laparoscopic procedure, requirement for reoperation within 30 days, wound infection, acute hydroceles and post-operative length of stay; 3) Long-term outcomes such as recurrent inguinal hernia, testicular atrophy and; 4) Cost of hospitalization will be compared between the open and laparoscopic groups.

Comparisons will be made in two groups of patients- patients with 1) unilateral hernias and 2) bilateral hernias and will last for 2 years. 102 patients in the unilateral arm and 50 patients in the bilateral arm will be randomized to each treatment group and each subject will be followed for up to 12 months following the surgical intervention. Two study evaluations by telephone (in addition to a single outpatient clinic visit already required as part of standard post-operative care) will be required of each research subject and his/her parent/guardian. The telephone evaluations will occur at 3 and 12 months following surgery. The standard post-operative clinic visit is scheduled at 2 weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than 3 years (36 months) at the time of surgery
2. Reducible inguinal hernia

Exclusion Criteria:

1. Concomitant need for other intraabdominal procedure
2. Prior inguinal hernia repair procedure
3. Hospitalization expected to be prolonged due to a concurrent illness actively being treated (e.g. congenital heart disease requiring surgical repair during the same hospitalization)
4. Liver Disease or contraindication to Tylenol, Midazolam, Fentanyl, or Marcaine.
5. Irreducible inguinal hernia, as determined in the operating room prior to randomization and incision.

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2007-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be total dose of acetaminophen administered for pain management. | 2 years

SECONDARY OUTCOMES:
Incidence of intraoperative complications: compromise of testicular vessels, perforation of abdominal viscera. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fizan Abdullah, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland